CLINICAL TRIAL: NCT01863693
Title: AN OBSERVATIONAL STUDY OF AVASTIN® (BEVACIZUMAB) AS FIRST LINE THERAPY IN PATIENTS WITH ADVANCED OVARIAN CANCER
Brief Title: An Observational Study of Avastin (Bevacizumab) in Combination With Chemotherapy as First-Line Treatment in Patients With Advanced Ovarian Cancer (OSCAR 1)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28570
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, prospective, observational study will evaluate the safety and efficacy of Avastin (bevacizumab) in combination with chemotherapy as first-line treatment in patients with advanced epithelial ovarian, fallopian tube or primary peritoneal cancer in routine clinical practice. Eligible patients will be followed for approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Advanced (FIGO stages IIIB, IIIC and IV) epithelial ovarian, fallopian tube or primary peritoneal cancer not previously treated with chemotherapy
* Initiating Avastin in combination with chemotherapy

Exclusion Criteria:

* Contraindications, warnings and precautions for use as specified in the Avastin Summary of Product Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced (FIGO stages IIIB, IIIC and IV) epithelial ovarian, fallopian tube, or primary peritoneal cancer undergoing first-line treatment with chemotherapy and Avastin
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival, defined as time from first administration of first-line therapy to documented disease progression | approximately 6 years
Safety: Incidence of adverse events | approximately 6 years

SECONDARY OUTCOMES:
Overall survival, defined as time from first administration of first-line therapy to documented death | approximately 6 years
Objective response rate, defined as percentage of patients with complete or partial response according to local assessments | approximately 6 years
Quality of life: EQ-5D/EORTC questionnaires | approximately 6 years
Dosage/schedule/duration of Avastin therapy | approximately 6 years
Composition of first-line chemotherapy regimens: drugs/dosage/duration | approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United Kingdom (30):
  - Royal United Hospital; Oncology Department, Bath
  - City Hospital, Birmingham
  - Bradford Royal Infirmary; Oncology Department, Bradford
  - Bristol Haematology and Oncology Centre, Bristol
  - Queen's Hospital; Oncology Department, Burton-on-Trent
  - Essex County Hospital, Colchester
  - Eastborne District General Hospital, Eastbourne
  - Wonford Hospital; Oncology Department, Exeter
  - Royal Surrey County Hospital, Guildford
  - Ipswich Hospital, Ipswich
  - Airedale General Hospital; Research Office Ward 12, Keighley
  - St James University Hospital, Leeds
  - Royal Marsden Hospital - London, London
  - Maidstone Hospital; Kent Oncology Centre, Maidstone
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - The James Cook University Hospital, Middlesbrough
  - Mount Vernon Hospital, Middlesex
  - St Mary's Hospital, Newport
  - City Campus; Academic Unit of Oncology, Nottingham
  - Queen Alexandra Hospital; Portsmouth Haematology & Oncology Centre, Level B, Portsmouth
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Southampton General Hospital, Southampton
  - City General Hospital, Stoke-on-Trent
  - The Royal Marsden Hospital, Sutton
  - Singleton Hospital; Oncology, Swansea
  - Torbay Hospital; Oncology Department, Torquay
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital; Deansley Centre, Wolverhampton
  - The York Hospital, York

REFERENCES:
- [Derived] Hall M, Bertelli G, Li L, Green C, Chan S, Yeoh CC, Hasan J, Jones R, Ograbek A, Perren TJ. Role of front-line bevacizumab in advanced ovarian cancer: the OSCAR study. Int J Gynecol Cancer. 2020 Feb;30(2):213-220. doi: 10.1136/ijgc-2019-000512. Epub 2019 Nov 27. PMID 31780570